CLINICAL TRIAL: NCT01537497
Title: Phase 1 Four-Arm Parallel Group, Placebo-Controlled Study To Evaluate The Effects Of Single Doses Of PF- 05175157 At Three Dose Levels On Pharmacodynamic And Metabolic Parameters In Healthy Volunteers
Brief Title: A Study To Evaluate The Effects Of PF-05175157 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1731013
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Phase 1; Single Doses; Pharmacodynamics; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100 mg PF-05175157 (Experimental): The chance of receiving 100 mg, 250 mg, 600 mg or placebo will be randomized.
  Interventions: Drug: PF-05175157
- 250 mg PF-05175157 (Experimental): The chance of receiving 100 mg, 250 mg, 600 mg or placebo will be randomized.
  Interventions: Drug: PF-05175157
- 600 mg PF-05175157 (Experimental): The chance of receiving 100 mg, 250 mg, 600 mg or placebo will be randomized.
  Interventions: Drug: PF-05175157
- Placebo (Placebo Comparator): The chance of receiving 100 mg, 250 mg, 600 mg or placebo will be randomized.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05175157 — One single oral dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM.
  Arms: 100 mg PF-05175157
Drug: PF-05175157 — One single oral dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM.
  Arms: 250 mg PF-05175157
Drug: PF-05175157 — One single oral dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM.
  Arms: 600 mg PF-05175157
Drug: Placebo — One single oral dose of placebo will be administered as a powder-in-capsule in the fasting state in the AM.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate pharmacodynamics of single oral doses of PF-05175157 in a dose-dependent fashion in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests. In addition, subjects must have normal pulmonary function tests and normal ocular findings.
* Women must be of non-childbearing potential.
* Body Mass Index (BMI) of 19.5 35.5 kg/m2, and a total body weight of > 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies and seasonal allergies at time of dosing).
* Evidence or history of any chronic ongoing or current pulmonary disease.
* History of smoking in the past 5 years or history or evidence of habitual use of other (non smoked) tobacco or nicotine-containing products within 3 months of Screening or positive cotinine test at Screening or Day -7.
* Active ocular disease including infection, glaucoma, seasonal allergies, dry eye symptoms or retinal/optic nerve disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Modulation of carbohydrate and lipid metabolism | 24 hours

SECONDARY OUTCOMES:
Cmax of PF-05175157 after single oral doses | 24 hours
Tmax of PF-05175157 after single oral doses | 24 hours
Area under the curve (AUC) of PF-05175157 after single oral doses | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731013&StudyName=A%20Study%20To%20Evaluate%20The%20Effects%20Of%20PF-05175157%20In%20Healthy%20Volunteers